CLINICAL TRIAL: NCT06790732
Title: The Effect of Preoperative Ultrasound-Guided Peri- Capsular Nerve Group Block on Postoperative Analgesia After Shoulder Arthroscopic Surgery
Brief Title: Preoperative Ultrasound-Guided Peri- Capsular Nerve Group Block on Postoperative Analgesia After Shoulder Arthroscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Kareem Ayman Khattab, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MS117/3/23
Record Dates: First submitted 2025-01-18; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Preoperative; Ultrasound-Guided; PeriCapsular Nerve Group Block; Postoperative Analgesia; Shoulder Arthroscopic Surgery
MeSH Terms: interventions — Sodium Chloride; Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Patients received sham PENG block (just 1mL saline).
  Interventions: Drug: Saline
- PeriCapsular Nerve Group Block (PENG) Group (Experimental): Patients received real PENG block (15 mL of bupivacaine 0.25% +0.2mg/mL dexamethasone).
  Interventions: Drug: Bupivacaine + Dexamethasone

INTERVENTIONS:
Drug: Saline — Patients received sham PENG block (just 1mL saline).
  Arms: Control Group
Drug: Bupivacaine + Dexamethasone — Patients received real PENG block (15 mL of bupivacaine 0.25% +0.2mg/mL dexamethasone).
  Other Names: PeriCapsular Nerve Group Block (PENG)
  Arms: PeriCapsular Nerve Group Block (PENG) Group

SUMMARY:
This study aimed to evaluate the analgesic efficacy of preoperative ultrasound-guided peri-capsular nerve group block (PENG) on postoperative analgesia after shoulder arthroscopic surgery.

DETAILED DESCRIPTION:
Postoperative pain control after shoulder surgery is challenging, and poor pain management is invariably reflected in poor outcomes, with longer hospitalization and recovery time. The difﬁculty in reducing pain due to the complexity of shoulder innervation leads to conducting studies to explore selective axillary nerve blocks with a posterior approach or from the axillae.

The peri-capsular nerve group (PENG) block is a regional anesthetic technique. It can be effectively and safely applied under ultrasound guidance in shoulder surgery cases for postoperative analgesia. It targets only the sensory branches and not the posterior mechanoreceptors; there is a potential motor-sparing effect which is desirable for better physical therapy, and earlier discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 65 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I-III.
* Scheduled for unilateral shoulder arthroscopic surgery.

Exclusion Criteria:

* Patient refusal.
* Known hypersensitivity to local anesthetics.
* Body mass index> 35 kg /m2.
* Uncooperative or psychiatric patients.
* Infection at the injection site.
* Coagulation disorder.
* Major cardiac, renal, or hepatic diseases.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Time to the first request of rescue analgesia | 24 hours postoperatively
  Time to the first request of rescue analgesia was recorded from the end of the surgery till first dose of morphine administrated.

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  The degree of pain was assessed using the Numerical Rating Scale (NRS) Pain score (metric score from 0 to 10 where 0 = no pain and 10 = maximal pain). NRS was recorded at PACU and 2, 4, 6, 8, 12, 16, 20, and 24 h postoperative.
Total morphine consumption | 24 hours postoperatively
  If patient numeric rating score was more than 3, patients received 3 mg morphine slowly intravenously. Morphine injection was repeated whenever required.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.